CLINICAL TRIAL: NCT00524706
Title: Phase I/II Study of S-1, Oral Leucovorin, and Oxaliplatin Combination Therapy (SOL) in Patients With Untreated Metastatic Colorectal Cancer
Brief Title: Phase I/II Study of SOL for Untreated Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shizuoka Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCC-07-01
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Cancer
Keywords: S-1; oral fluoropyrimidine; tegafur; Gimeracil; Oteracil Potassium; Leucovorin; Calcium Folinate; Oxaliplatin; L-OHP; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: S-1, oral Leucovorin, Oxaliplatin

SUMMARY:
Introduction:

S-1 is promising drug which could replace 5-fluorouracil plus l-leucovorin (5-FU/l-LV) in treatment of advanced colorectal cancer.

Phase I/II study of S-1 plus Oxaliplatin (SOX) demonstrated its promising activity with acceptable toxicity as first-line chemotherapy in patients with untreated metastatic colorectal cancer and S-1 showed equivalent possibility to 5-FU/l-LV. On the other hand, phase I/II study of S-1 plus oral Leucovorin (S-1/LV) demonstrated that this regimen had enhanced efficacy in comparison with S-1 alone. From these results, it was expected that S-1/LV plus Oxaliplatin (SOL) would be more effective than SOX.

Therefore, phase I/II study of SOL combination therapy was planned.

Purpose A dose-finding study of S-1/LV plus Oxaliplatin (SOL) was planned to determine the recommended dose (RD), and to assess the response rate (RR) in patients with untreated metastatic colorectal cancer. The primary endpoints of the phase I portion are determination of the RD of SOL, and safety.

The phase II portion of this study was aimed to assess the RR of SOL.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Adequate oral intake.
* Histologically proved adenocarcinoma (colorectal cancer).
* Unresectable, recurrent and advanced colorectal cancer.
* At least 4 weeks since prior major surgery
* Age: 20 - 74 at enrollment.
* Performance Status (Eastern Cooperative Oncology Group [ECOG] scale): 0 - 2.
* No prior treatment (ex. radiation therapy, chemotherapy, hormonal therapy) to advanced disease. Patients who received adjuvant chemotherapy more than 180 days before enrollment can be allowed but those who received S-1 or Oxaliplatin containing treatment shall be excluded.
* Proved presence of measurable lesions within 30 days before enrollment.
* Patients with the following function of bone marrow, liver and kidney based on the laboratory values measured within 15 days before enrollment.

  * Hemoglobin >_ 9.0g/dL
  * WBC: LLN - 12,000/mm3
  * Absolute granulocyte count >_ 1,500/mm3
  * Platelets >_ 100,000/mm3
  * Total Bilirubin <_ 1.5mg/dL
  * AST(GOT) and ALT(GPT) <_ 100U/L
  * ALP <_ 600U/L
  * Creatinine <_ 1.0mg/dl
* Expected to survive more than 90 days after enrollment.

Exclusion Criteria:

* Patients who not received S-1 and Oxaliplatin as neoadjuvant or adjuvant chemotherapies before enrollment.
* Contraindication to S-1, and serious hypersensitivity to oral Leucovorin.
* No other concurrent investigational therapy.
* Patients did who not received blood transfusion and hematogenesis stimulating agents (ex. Granulocyte-Colony Stimulating Factor).
* Serious drug hypersensitivity.
* Prior history of peripheral neuropathy.
* Marked infection or inflammation (ex. patients with a fever of 38.0 degrees or higher).
* Poorly-controlled diabetes, hypertension or hypercalcemia.
* Severe (inpatient care is needed) arrhythmia, heart disease or its history.
* Severe (inpatient care is needed) lung disease (ex. interstitial pneumonia or pulmonary fibrosis).
* Psychiatric disorder requiring to receive treatment with antipsychotic drug.
* Fresh bleeding from the gastrointestinal tract.
* Requiring to drainage massive ascites, pleural effusion retention or pericardial fluid.
* Extensive bone metastasis.
* Clinically suspicious brain metastasis or brain metastasis.
* Diarrhea (watery diarrhea).
* Simultaneously active double cancer.
* Pregnancy or nursing female patients and possibility (intent) to bear baby. Male patients with intent to impregnate.
* Other patients evaluated to be inadequate to participate in the study by (sub) investigators.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-08; Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Determine the RD of S-1, Leucovorin, and Oxaliplatin in phase I setting | During 2 cycles
Evaluate the response rate of S-1, Leucovorin, and Oxaliplatin with recommended dose in phase II | During chemotherapy

SECONDARY OUTCOMES:
Phase I - Safety - Pharmacokinetic drug-drug interaction - Response rate - Time to treatment failure (TTF) - Progression free survival (PFS) - Overall survival (OS)
Phase II - Safety - Time to treatment failure (TTF) - Progression free survival (PFS) - Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Narikazu Boku, MD, Principal Investigator — Shizuoka Cancer Cener, Division of Gastrointestinal Oncology
Locations (1):
- Shizuoka Cancer Center, Shizuoka, Japan